CLINICAL TRIAL: NCT05794646
Title: Community Intervention to Eliminate HCV Among People Who Use Drugs. Implementation Study in the Cities of Paris, Marseille, Lyon and Fort-de-France, France.
Brief Title: Community Intervention to Eliminate HCV Among People Who Use Drugs.
Acronym: ICONE2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 0336s ICONE 2
Record Dates: First submitted 2023-03-06; First posted 2023-04-03 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: HCV; Substance Use Disorders
Keywords: Hepatitis C Virus; mental health; RDS; peers; Test and Treat; People who use drugs
MeSH Terms: conditions — Substance-Related Disorders; Hepatitis C; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This type 2 hybrid 'effectiveness-implementation' study makes it possible to simultaneously evaluate the efficiency of the model on clinical criteria of HCV cure, and its feasibility by measuring the potential obstacles and the relevance of its implementation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Other): Community-based intervention with screening and treatment initiation for HCV elimination among PWUD
  Interventions: Other: Hybrid effectiveness-implementation study type 2

INTERVENTIONS:
Other: Hybrid effectiveness-implementation study type 2 — Diagnosis of hepatitis C; Assessment of hepatic fibrosis; Treatment of hepatitis C; Assessment of psychological disorders and treatment or referral.

SUMMARY:
The goal of this interventional study is twofold with the evaluation of the feasibility and potential usefulness of an implementation strategy, and the efficiency of a community-based model of mass screening and immediate treatment of hepatitis C among People Who Use Drugs (PWUD) in three major cities in mainland France (Paris, Lyon and Marseille) and in one overseas city (Fort-de-France). The investigators will also describe the psychological and infectious comorbidities of drug users, determine the stages of the HCV (Hepatitis C Virus), HBV (Hepatitis B Virus), HIV (Human Immunodeficiency Virus) care cascade, and analyze the factors associated with HCV treatment failure. A qualitative study will investigate the acceptability of the RDS model.

Participants will be screened in an out of bound research center and receive appropriate treatment for infectious, addictological and psychiatric troubles. They will receive coupons to give to their peers for them to participate in the study.

Researchers will also compare the acceptability of referral to psychiatric care directly at the research site (intervention group) with that of referral directly to a city facility (control group).

DETAILED DESCRIPTION:
Current state of knowledge:

In France, the prevalence of chronic hepatitis C in the general population was 0.3% in 2015. However, this prevalence is much higher in certain population subgroups. Thus PWUD are a population at risk of HCV infection (risky behaviors, sharing injection equipment).

In order to achieve the goal of eliminating hepatitis C by 2025 in France, three types of actions must be taken: developing off-premises screening strategies, improving access to treatment, and improving prevention. These actions correspond to micro-elimination practices.

Although there are many possible sites of care for PWUD, many PWUD do not attend the prevention and care system.

Despite the advent of new direct antiviral agents (DAAs) that cure infection in more than 95% of cases and the indication to treat all PWUDs, access to HCV treatment in this at-risk group remains low. Better control of HCV infection in high-risk groups such as PWUD would, beyond the individual benefit, greatly reduce the dynamics of the epidemic.

The prevalence of psychiatric disorders in the PWUD population, especially the most precarious, is high, with at least one characterized psychiatric disorder observed in 50% to 80% of situations. The existence of unrecognized and untreated psychiatric disorders in these subjects is a factor of lesser access to somatic care, in particular to HCV care. Therefore, optimizing access to HCV care in the PWUD population requires the identification and appropriate management of psychiatric pathologies in these individuals.

Research Hypothesis:

The investigators hypothesize that the Respondent Driven Sampling (RDS) recruitment technique and the community-based approach can be implemented in large urban areas and legally allow for psychiatric support, often necessary in this vulnerable population.

This study will also make it possible to estimate the size of the different populations of drug users in 4 large cities in France, one of which is overseas, in which the local specificities in terms of drug use but also of comorbidities will have to be studied (Capture/recapture).

In addition, the use of this recruitment technique coupled with the involvement of peers, will make it possible to define the different drug uses in the user population in the major cities of metropolitan France and in Fort-de-France. This information obtained from a population of hidden users is important and complementary to the results of the studies carried out in center for taking care of addiction problems (CSAPA) and support centres for the reduction of drug-related harms (CAARUD), by the ANRS (The French agency for AIDS and viral hepatitis research) 14059s Coquelicot study.

Furthermore, the investigators hypothesize that the multicentric implementation of this screening and treatment strategy will be facilitated by the use of a toolkit. This toolkit "ICONE" has been developed by the investigating team of the ANRS 95050 ICONE study.

Finally, the investigators hypothesize that the proposal to initiate psychiatric follow-up at the site of the RDS will have an effect on the insertion into city mental health care in the months following the RDS in PWUD with psychiatric comorbidities.

Principal objective:

The main objective is twofold with the evaluation of the feasibility and potential usefulness of an implementation strategy, and the efficiency of a community-based model of mass screening and immediate treatment of hepatitis C among PWUD in Paris, Marseille, Lyon and Fort-de-France.

Secondary objectives:

* Estimate the size of the PWUD population in the 4 cities;
* Determine the prevalence of chronic HCV infection in the PWUD population in the 4 cities;
* Estimate the steps in the retrospective HCV care cascade (positive HCV Rapid Diagnostic Test (RDT), known HCV status, previously initiated antiviral therapy, undetectable viral load) ;
* Determine the factors associated with hepatitis C treatment failure: defined as a detectable viral load 12 weeks after the end of treatment;
* Estimate the cost of our intervention for one PWUD screened and one PWUD cured of hepatitis C;
* Estimate the prevalence of HIV infection among PWUDs in the 4 cities;
* Estimate the steps in the retrospective care cascade of HIV infection (known HIV status, previously initiated antiviral treatment, undetectable viral load);
* Estimate the prevalence of chronic hepatitis B among PWUD in the 4 cities;
* Estimate the prevalence of sexually transmitted infections (STIs) (Syphilis, Gonorrhoea, Chlamydia) among PWUD in Fort-de-France;
* Describe the most frequent psychological comorbidities in the PWUD population in the 4 cities;
* Evaluate the effectiveness of peer-supported referral to infectious (HIV, HCV, HBV at all sites and STIs only in Fort-de-France), psychiatric and addictive care;
* To compare the acceptability of referral to psychiatric care directly at the research site (intervention group) with that of referral directly to a city facility (control group).

All of these objectives will be analyzed specifically in the sub-population of crack cocaine users.

Qualitative study objectives Evaluate the acceptability of the RDS model and the relevance of an implementation strategy.

Methodology:

Hybrid effectiveness-implementation study type 2, allowing to evaluate simultaneously the effectiveness of the model on clinical criteria of access to psychiatric, addictological and infectious diseases care, and its feasibility by measuring the levers and potential obstacles to its implementation.

For the qualitative part, the investigators will conduct 15 interviews per site, i.e. 60 semi-structured interviews with the PWUDs who participated in the RDS. The researchers will organize 1 focus group with the stakeholders of each site before and after the implementation of the RDS.

Intervention:

Recruitment of PWUDs will be done through an RDS method. Ten to fifteen "seeds" will be selected per city for their diversity and social network. They will be invited to the research site (temporary community care facility), participate in all study procedures, and then receive 2-3 coupons to recruit eligible peers. Participants will receive HCV/HIV/HBV screening, on-site HCV RNA testing, liver fibrosis measurement, rapid antiviral (HCV) treatment initiation, treatment monitoring, and risk and harm reduction tools related to their risky practices. Participants with an HIV and/or HBV positive RDT will be referred to infectious disease services and the referral will be assessed. An assessment of psychological disorders will be carried out by i) Quick Screening Tool (QST) questionnaire asked to all participants; ii) MINI questionnaire for participants with positive QST. In case of a positive MINI, psychiatric consultations will be offered on site (Paris and Fort-de-France) or participants will be referred to structures offering psychiatric care (Lyon, Marseille). The effectiveness of referral to psychiatric care between the two interventions will be compared. All RDS participants will be referred to permanent addiction facilities and this referral will be evaluated. Peers will be present at this unique facility and will accompany participants throughout their HCV treatment. A capture/recapture study, nested within the RDS, will provide a reliable estimate of the PWUD population in the Paris arrondissements covered by the RDS and the cities of Marseille, Lyon and Fort-de-France. The qualitative study will take place at all sites. Individual interviews for a total of 60 participants will be conducted, as well as focus groups with stakeholders in each site.

Statistical methods:

Categorical variables will be described in terms of numbers and percentages with their associated 95% confidence intervals calculated using the exact method. Comparisons will be carried out by Chi² or Fisher's exact tests. Continuous variables will be described in terms of numbers, median, range and interquartile range or mean, standard deviation, standard deviation of the mean and confidence interval. Comparisons will be carried out using Mann-Whitney or Student's t tests depending on the distribution of the variable. The estimation of the size of the drug user populations will use the method recommended by the WHO (World Health Organization) with the Lincoln-Peterson estimator. Missing data will be taken into account by adopting the most penalizing approach. Logistic regression models will be used to search for factors associated with treatment failure. Multivariate logistic regression models will be employed to compare the success of psychiatric referral between the two groups.

Anticipated schedule:

Expected start date of the research (opening of RDS): September 2023 Duration of inclusions: 3 or 4 months per site (not necessarily over the same period) Duration of participation per participant: 1 day to 9 months Total expected duration of research: 24 months Anticipated end date of the trial/research: September 2025

Timeline for follow-up of participants in the research:

Participants with HCV RNA positive at RDS will be followed until SVR12 from treatment initiation. Visits at S4, end of treatment and SVR12.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years;
* Person who uses drugs, defined as:
* Reported psychoactive substance use and
* Positive urine test for at least one of the following: heroin, amphetamines, cocaine, MDMA (methylenedioxymethamphetamine), ecstasy, or misused opioid medications (methadone, buprenorphine or opiates used for a reason other than its original prescription (effects seeking) or used in a way that does not comply with its marketing authorisation (injected, snorted, taken multiple times beyond the prescribed dosage)) ;
* Informed and signed consent

Exclusion criteria:

* Inability to understand the study;
* Being under guardianship, curatorship or mandate of future protection;
* Person participating in another research study with an exclusion period still in progress at the time of pre-inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of HCV cured PWUD participants (SVR12) among those with a positive HCV viral load at baseline | 12 weeks after the end of the 2 to 3 months HCV treatment
  Number of HCV cured PWUD participants, defined as SVR12, i.e. undetectable HCV RNA viral load in a veinous sample measured by quantitative PCR (polymerase chain reaction) 12 weeks after the end of the antiviral treatment; divided by the number of participants with a positive HCV viral load in a veinous sample at baseline.
Acceptability and relevance of the RDS and implementation strategy : a qualitative study | From before the RDS implementation until the end of the study, up to 2 years
  The investigators will use a socio-anthropological method to target the PWUD participating in the RDS as well as the workers in the places where the RDS will have started.
  In each study city, 15 semi-structured interviews will be conducted with PWUD who participated in the RDS. Participants who are not followed up in outreach structures will be over-represented to delve deeper into the pathways of these individuals.
  Two focus groups in each city will be carried-out (one before the implementation of the RDS and one at the end of the study), in order to collect their feelings on the use and relevance of the toolkit for the implementation of the RDS.
  The interviews and focus groups will be conducted using an interview grid that will be constructed to meet the objectives of the study. This grid will guide the investigators around different main themes: people's backgrounds, role of the facilitators, perception of RDS (understanding, acceptability, strengths and weaknesses).

SECONDARY OUTCOMES:
Number of PWUD in the arrondissements of Paris (neighborhoods involved in seed distribution), and the cities of Lyon, Marseille and Fort-de-France | At the end of the RDS
  Estimated Number of PWUD in the arrondissements of Paris (neighborhoods involved in seed distribution), and the cities of Lyon, Marseille and Fort-de-France
Proportion of participants with positive HCV RNA among all participants | At baseline
  Number of participants with a positive HCV RNA divided by the number of participants
Assessment of HCV cascade of care at inclusion : participants with a positive HCV RDT | At baseline
  Number of participants with a positive HCV RDT
Assessment of HCV cascade of care at inclusion : participants with known HCV status | At baseline
  Number of participants with known HCV status (declarative) among participants with a positive HCV RDT
Assessment of HCV cascade of care at inclusion : participants who were treated for HCV | At baseline
  Number of participants who were treated for HCV (self-reported) among participants with known HCV status
Assessment of HCV cascade of care at inclusion : participants with known chronic hepatitis C status and undetectable HCV RNA | At baseline
  Number of participants with known chronic hepatitis C status and undetectable HCV RNA among participants who were treated for HCV
HCV treatment failure defined as detectable viral load 12 weeks after HCV treatment completion | 12 weeks after the end of the 2 to 3 months HCV treatment
  HCV treatment failure defined as detectable HCV RNA viral load measured in a veinous sample by quantitative PCR 12 weeks after the end of the antiviral treatment
Cost of the intervention per screened participant | Through study completion, an expected time frame of 2 years
  All costs of the intervention divided by the number of participants screened
Cost of the intervention per participant cured of hepatitis C | Through study completion, an expected time frame of 2 years
  All costs of the intervention divided by the number of participants cured of hepatitis C
Proportion of participants with a positive HIV RDT among participants | At baseline
  Number of participants with a positive HIV RDT divided by the number of participants
HIV care cascade assessment at inclusion : participants with known HIV status | At baseline
  Number of participants with known HIV status
HIV care cascade assessment at inclusion : HIV-positive participants on antiretroviral therapy | At baseline
  Number of HIV-positive participants on antiretroviral therapy among participants with known HIV status
HIV care cascade assessment at inclusion : participants on effective antiretroviral therapy | At baseline
  Number of participants on effective antiretroviral therapy (HIV RNA < 50 copies/ml) among HIV-positive participants on antiretroviral therapy
Proportion of participants with detectable HBsAg | At baseline
  Number of participants with detectable HBsAg divided by the number of participants
Proportion of participants in Fort-de-France with a positive PCR for gonorrhea | At baseline
  Number of participants in Fort-de-France with a positive PCR for gonorrhea divided by the number of participants in Fort-de-France
Proportion of participants in Fort-de-France with a positive PCR for chlamydia | At baseline
  Number of participants in Fort-de-France with a positive PCR for chlamydia divided by the number of participants in Fort-de-France
Proportion of participants in Fort-de-France with a positive test for syphilis | At baseline
  Number of participants in Fort-de-France with a positive test for syphilis divided by the number of participants in Fort-de-France
Prevalence of psychological pathologies | At baseline
  Prevalence of psychological pathologies diagnosed by the MINI questionnaire (nurse trained beforehand notably on the psychosis module) with the use of 3 modules: Major depressive episode, psychotic disorders and suicidal risk following the positive QST questionnaire
Success of infectious diseases referral | At 6 months
  Proportion of participants referred to an infectious diseases structure who went to their consultation
Success of addictological referral | At 6 months
  Proportion of participants referred to an addictological structure who went to their consultation
Success of psychiatric referral at 3 months | At 3 months
  Proportion of participants referred to a psychiatric structure in the city who went to their consultation
Success of psychiatric referral at 6 months | At 6 months
  Proportion of participants referred to a psychiatric structure in the city who went to their consultation

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Donnadieu, PhD, Principal Investigator — PCCEI
Locations (4):
- France (3):
  - Lyon, Lyon, Auvergne-Rhône-Alpes
  - Marseille, Marseille, PACA
  - Paris, Paris, Île-de-France Region
- Martinique, Fort-de-France, Martinique, Martinique

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data
Time Frame: After publication and for 15 years.
Access Criteria: Open to anyone at https://recherche.data.gouv.fr/